CLINICAL TRIAL: NCT05784792
Title: Clinical and Surgical Outcomes of Total Thyroidectomy in Basedow's Disease: the Effect of Lugol Solution
Acronym: BALU
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Maurizio Iacobone, MD, FEBS (Endocrine Surgery), Associate Professor, Head in Chief of Endocrine Surgery Unit of Padua University Hospital, Italy, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPd39962
Record Dates: First submitted 2023-01-27; First posted 2023-03-27 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Basedow Disease
Keywords: Lugol Solution; Total Thyroidectomy
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Intervention Model Description: Case-Control study
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lugol - (No Intervention): No pre-operative Lugol Solution preparation
- Lugol + (Active Comparator): Pre-operative Lugol preparation (10 drops per day orally three times a day for 7 days for an amount of 10,5 ml of Lugol solution that contains 1,68 gr of Iodine).
  Interventions: Other: Lugol -

INTERVENTIONS:
Other: Lugol - — Patients that undergo total thyroidectomy without Lugol solution pretreatment
  Arms: Lugol +

SUMMARY:
Preoperative preparation of patient with Basedow's disease is crucial to avoid severe thyrotoxicosis resulting from leakage of thyroid hormone into the circulation at the time of surgery. Moreover, hyperthyroidism-related hypervascularization and tissue fragility caused by Basedow's disease thyroiditis may cause intraoperative bleeding that can reduce the visualization and preservation of parathyroid glands and laryngeal nerves with subsequent higher risk of related morbidity including neck hematoma, hypoparathyroidism and vocal cords paresis. Although some endocrine surgeons administer before surgery Lugol solution to decrease thyroid gland vascularity in Basedow's disease, there is still not an agreement on its effectiveness.

The aims of the present trial are to evaluate the impact of pre-operative short-term Lugol solution treatment (7 days) on surgical outcomes through modification of thyroid vascularity and surgical related morbidity, in patients with Basedow's disease.

DETAILED DESCRIPTION:
The study will investigate the effects of Lugol solution treatment before surgery on thyroid vascularity and tissue fragility in patients with Basedow's disease, and if these changes are associated or not with different surgical outcomes.

Hyperthyroidism is associated with hemodynamic changes, decreasing peripheral resistance that are related to both direct cardio-stimulatory effects of thyroid hormone. Preoperative preparation of the patient is crucial to avoid intra-operative or postoperative thyroid storms and to decrease the vascularity of the gland.

Inorganic iodide (Lugol solution) decreases the synthesis of thyroid hormone and release of hormone from the thyroid in the short term. Iodine also seems to reduce thyroid cellularity and vascularity and therefore is used in the preparation of patients for thyroidectomy. This effect transiently blocks thyroid hormone generation, with thyroid hormone synthesis recovering in few days.

On this matter doppler techniques seem to be the best method to evaluate blood flow in the thyroid gland.

Thyroid vascularity in Basedow's disease patients can be evaluated by monitoring CD-34 and CD-31 expression using immunohistochemistry. The vascular density of different tissues has been assessed by counting vessels labeled using immunohistochemistry with antibodies against different endothelial markers on paraffin-embedded sections. Antibodies that are most commonly used are directed against the endothelial antigens factor eight-related antigen, CD-31 (platelet endothelial cell adhesion molecule), CD-34. CD-34 is the most sensitive and specific marker currently available for the detection of angiogenesis. The use of these markers reflects total vascular density.

Moreover some authors showed that iodide inhibits vascular endothelial growth factor (VEGF) expression in cultured human thyroid follicles, and, consequently, they suggest that pro-angiogenic and anti-angiogenic factors may at least partly account for the iodide-induced decrease in thyroid blood flow. Cross-talk between angiogenesis and inflammation has also been reported. T cells can deliver VEGF to inflammatory sites and VEGF can augment pro-inflammatory T cell differentiation and promote angiogenesis.

So the detection of VEGF could be useful in the demonstration of Lugol effect on pretreated patients.

Investigators hypothesize that Lugol solution might act through different mechanisms. It probably decreases both angiogenic stimuli and blood flow in Basedow's disease. Decreased angiogenesis and blood flow resulted in a significantly decreased number of visible vessels. Therefore, it is reasonable to think that increased vascular density could reflect increased angiogenic input to this disease. Lugol solution could also act directly to vessels wall, changing arteries and veins lumen.

These modifications could cause a reduction of intra-operative bleeding that could allow better visualization and preservation of the surrounding nerves, vasculature, and parathyroid glands and so better surgical and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Basedow disease candidate to total thyroidectomy
* age>18 years

Exclusion Criteria:

* age<18 years;
* presence of solitary toxic nodule
* fine-needle aspiration biopsy result indicating cancer or suspicious cytology
* anticoagulant usage or coagulation disorders
* a previous thyroid operation
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2024-04-26 (Estimated)

PRIMARY OUTCOMES:
Intra and post-operative blood loss (mL). | Intra and post-operative bleeding (1st and 2nd day after surgery)
  Blood loss volume (mL) as the amount of blood in the suction bottle and that absorbed by gauzes used during surgery was measured (volume calculated from the difference between dry gauzes weight and soaked gauzes weight). Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).

SECONDARY OUTCOMES:
Post-operative laryngeal nerves palsy. | Laryngeal ultrasound on 1st and 2nd day and indirect laryngoscopy in case of dysphonia
  Evaluation of vocal cords disfunction. Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Intra and post-operative thyrotoxicosis. | During surgery and on 1st and 2nd day after surgery
  Heart rate > 120 b/min detected during surgery or during post-operative hospital days. Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Post-operative hypocalcemia (hypoparathyroidism, hungry bone syndrome). | Blood sample on 1st and 2nd day after surgery.
  serum calcium level less than 2,00 (8 mg/dl), with serum PTH inappropriately low (<10 pg/mL). Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).

OTHER OUTCOMES:
Change of ultrasound thyroid vascularization: blood flow velocity (v) variation (mm/sec). | Thyroid US doppler data: 7 days before surgery and the day before surgery (after 1 week).
  US doppler of 4 thyroid arteries: blood flow velocity (v) (mm/sec) of the four main thyroid arteries, sampled near their entrance into the gland. Mean values for each artery is than calculated. Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of ultrasound thyroid vascularization: resistance index (RI) variation. | Thyroid US doppler data: 7 days before surgery and the day before surgery (after 1 week).
  US doppler of 4 thyroid arteries: resistance index (RI) of the four main thyroid arteries, sampled near their entrance into the gland. It is the ratio between (peack systolic velocity-end diastolic velocity)/peack systolic velocity. Mean values for each artery is than calculated. Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of ultrasound thyroid vascularization: pulsatility index (PI) variation | Thyroid US doppler data: 7 days before surgery and the day before surgery (after 1 week).
  US doppler of 4 thyroid arteries: pulstility index (PI) of the four main thyroid arteries, sampled near their entrance into the gland. It is the ratio between (peack systolic velocity-end diastolic velocity)/mean velocity. Mean values for each artery is than calculated. Evaluation of differences in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of US thyroid volume (mL). | Thyroid US doppler data: 7 days before surgery and the day before surgery (after 1 week). Intra-operative thyroid volume detection (the day of surgery).
  Thyroid volume recorded through ultrasound (mL). It is also recorded directly after gland excision in the operating room (measuring the modification of the water volume inside a bowl after having dip the excised gland in the water bowl itself). Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of thyroid tissue: immunohistochemical evaluation of thyroid tissue mean vessels density. | Post-operative pathological and immunoistochemical data recorded (in 30 days after surgery).
  Thyroid vascularity evaluated through data recorded by hematoxylin and eosin sections and additional sections immunostained for CD-34 and CD-31. Section are scanned and mean vessels density is calculated by a specific softwear that recognizes CD31 and CD34 endothelial expression (specific colour expressed). The final count is then made by the softwear itself that through a machine learning method gives the section vessels total number and roe representative area mean vessels density. Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of thyroid vascularization stimuli: VEGF levels variation (pg/mL). | Blood samples: 7 days before surgery and the day before surgery (after 1 week).
  Thyroid vascularity evaluated through variation of VEGF plasmatic concentration (pg/mL) before and after Lugol solution assumption (when administrated). Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of thyroid function and biochemical data: FT3 and FT4 variation (pmol/L). | Blood samples: 7 days before surgery and the day before surgery (after 1 week).
  Serum FT3 and FT4 (pmol/L) levels variation before and after Lugol solution assumption (when administrated). Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of thyroid function and biochemical data: TSH variation (mIU/L). | Blood samples: 7 days before surgery and the day before surgery (after 1 week).
  Serum TSH (mIU/L) levels variation before and after Lugol solution assumption (when administrated). Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).
Change of thyroid function and biochemical data: Ab anti TG, Ab anti TPO, Ab anti TSH variation (U/L). | Blood samples: 7 days before surgery and the day before surgery (after 1 week).
  Serum Ab anti TG, Ab anti TPO, Ab anti TSH levels (U/L) variation before and after Lugol solution assumption (when administrated). Evaluation of differences (if any) in this outcome in the two groups of the study (Lugol assumption/no Lugol assumption).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Iacobone, Prof, Study Director — University of Padova
Locations (1):
- Azienda Università di Padova, Endocrine Surgery Unit, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hope N, Kelly A. Pre-Operative Lugol's Iodine Treatment in the Management of Patients Undergoing Thyroidectomy for Graves' Disease: A Review of the Literature. Eur Thyroid J. 2017 Feb;6(1):20-25. doi: 10.1159/000450976. Epub 2016 Nov 22. PMID 28611944
- [Result] Erbil Y, Ozluk Y, Giris M, Salmaslioglu A, Issever H, Barbaros U, Kapran Y, Ozarmagan S, Tezelman S. Effect of lugol solution on thyroid gland blood flow and microvessel density in the patients with Graves' disease. J Clin Endocrinol Metab. 2007 Jun;92(6):2182-9. doi: 10.1210/jc.2007-0229. Epub 2007 Mar 27. PMID 17389702
- [Result] Yilmaz Y, Kamer KE, Ureyen O, Sari E, Acar T, Karahalli O. The effect of preoperative Lugol's iodine on intraoperative bleeding in patients with hyperthyroidism. Ann Med Surg (Lond). 2016 Jun 16;9:53-7. doi: 10.1016/j.amsu.2016.06.002. eCollection 2016 Aug. PMID 27408715
- [Result] Shinall MC Jr, Broome JT, Nookala R, Shinall JB, Kiernan C, Parks L 3rd, Solorzano CC. Total thyroidectomy for Graves' disease: compliance with American Thyroid Association guidelines may not always be necessary. Surgery. 2013 Nov;154(5):1009-15. doi: 10.1016/j.surg.2013.04.064. Epub 2013 Sep 26. PMID 24075271
- [Result] Huang SM, Liao WT, Lin CF, Sun HS, Chow NH. Effectiveness and Mechanism of Preoperative Lugol Solution for Reducing Thyroid Blood Flow in Patients with Euthyroid Graves' Disease. World J Surg. 2016 Mar;40(3):505-9. doi: 10.1007/s00268-015-3298-8. PMID 26546192
- [Result] Yabuta T, Ito Y, Hirokawa M, Fukushima M, Inoue H, Tomoda C, Higashiyama T, Kihara M, Uruno T, Takamura Y, Kobayashi K, Miya A, Matsuzuka F, Miyauchi A. Preoperative administration of excess iodide increases thyroid volume of patients with Graves' disease. Endocr J. 2009;56(3):371-5. doi: 10.1507/endocrj.k08e-240. Epub 2009 Jan 9. PMID 19139595
- [Result] Smith TJ, Hegedus L. Graves' Disease. N Engl J Med. 2016 Oct 20;375(16):1552-1565. doi: 10.1056/NEJMra1510030. No abstract available. PMID 27797318
- [Result] Ansaldo GL, Pretolesi F, Varaldo E, Meola C, Minuto M, Borgonovo G, Derchi LE, Torre GC. Doppler evaluation of intrathyroid arterial resistances during preoperative treatment with Lugol's iodide solution in patients with diffuse toxic goiter. J Am Coll Surg. 2000 Dec;191(6):607-12. doi: 10.1016/s1072-7515(00)00755-9. PMID 11129808
- [Result] Erbil Y, Giris M, Salmaslioglu A, Ozluk Y, Barbaros U, Yanik BT, Kapran Y, Abbasoglu SD, Ozarmagan S. The effect of anti-thyroid drug treatment duration on thyroid gland microvessel density and intraoperative blood loss in patients with Graves' disease. Surgery. 2008 Feb;143(2):216-25. doi: 10.1016/j.surg.2007.07.036. Epub 2007 Dec 21. PMID 18242338
- [Derived] Schiavone D, Crimi F, Cabrelle G, Pennelli G, Sacchi D, Mian C, Torresan F, Iacobone M. Role of Lugol solution before total thyroidectomy for Graves' disease: randomized clinical trial. Br J Surg. 2024 Aug 2;111(8):znae196. doi: 10.1093/bjs/znae196. PMID 39129619